CLINICAL TRIAL: NCT06571292
Title: Effectiveness of Dose-intensity Therapy in Post-stroke Upper Limb Rehabilitation: an Occupational Therapy Approach
Brief Title: Effectiveness of Intensive Training in Upper Limb Rehabilitation After Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Enrique Villa Berges, PhD Principal investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University Zaragoza
Record Dates: First submitted 2024-07-11; First posted 2024-08-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Stroke; intensive training; upper limb; occupational therapy
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The principal investigator will not carry out any intervention or outcome evaluation.
  Both the principal investigator and the investigators of the interventions will be blinded to the data of the measurements that have been taken, and must leave the room during the assessment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): The control group will be trained with robotic exoskeleton for upper limbs and task specific training, 3 sessions per week for 4 weeks, for 1 hour per day.
  Interventions: Device: Intensive training with robotic exoskeleton for upper limbs; Device: Task specific training
- Intensive group (Experimental): The intensive group will be trained with robotic exoskeleton for upper limbs and task specific training, 5 sessions per week for 4 weeks, for 2 hours per day.
  Interventions: Device: Intensive training with robotic exoskeleton for upper limbs; Device: Task specific training

INTERVENTIONS:
Device: Intensive training with robotic exoskeleton for upper limbs — Both groups will be trained with robotic exoskeleton for upper limbs and task specific training.
Device: Task specific training — Both groups will be trained with robotic exoskeleton for upper limbs and task specific training.

SUMMARY:
The aim of the study is to analyse the effect of intensive training on upper limb function in stroke patients.

16 stroke patients were randomly divided into two groups: the intensive group and the control group.

The control group will be trained with robotic exoskeleton for upper limbs and task specific training, 3 sessions per week for 4 weeks, for 1 hour per day.

The intensive group will do robotic exoskeleton for upper limbs and task specific training, 5 sessions a week for 4 weeks, for 2 hours a day.

DETAILED DESCRIPTION:
Abtract

Aim: The aim of the study is to analyze the effect of intensive training on upper limb function in stroke patients.

Methods: The control group will be trained with robotic exoskeleton for upper limbs and task specific training, 3 sessions per week for 4 weeks, for 1 hour per day.

The intensive group will do robotic exoskeleton for upper limbs and task specific training, 5 sessions a week for 4 weeks, for 2 hours a day. The primary outcome measure include is the Fugl Meyer Assessment (FMA).Secondary measures include the Box and Blocks Test (BBT), dynamometer, Motor Activity Log (MAL), Stroke Impact Scale (SIS), Functional Independence Measure (FIM) and Canadian Occupational Performance Measure (COPM).

Assessments occur at baseline, after 4 weeks of intervention, and at 1 month after intervention commencement. Analysis will be intention to treat using a generalised linear mixed model to report estimated mean differences in scores between the two groups at each timepoint with 95% confidence Interval and value p.

Hypothesis: If an intensive training programme is effective in improving upper limb motor function, its implementation for clinical practice could be beneficial for improving upper limb motor function and quality of life in people who have suffered a stroke.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with stroke (ischaemic or haemorrhagic).
* Patients in a subacute or chronic state.
* Patients must be over 18 years of age and under 80 years of age.
* Patients with impaired functionality of the upper limb.

Exclusion Criteria:

* Persons diagnosed with other pathologies, other than those indicated in the inclusion criteria.
* Mini-Mental State Examination (MMSE), the minimum score to be achieved will be 22 points.
* Severe difficulties in understanding language (aphasia).
* Behavioural or behavioural disturbance.
* Treatment with botulinum toxin 3 months prior to the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assesment (FMA) | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement
  Primary Outcome Measure. It is a scale where the area of assessment includes ADLs, functional mobility and pain. ICF Domain, Body Function.Minimal Detectable Change (MDC) FMA = 5.2 points for the Upper Extremity portion of the assessment

SECONDARY OUTCOMES:
Box and Blocks Test (BBT) | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures.Assesses unilateral gross manipulative skills.ICF Domain Activity.Minimal Detectable Change (MDC)MDC: 5.5 blocks per minute
Dynamometer | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures.A quantitative and objective measure of isometric muscular strength of the hand and forearm. ICF Domain Body Structure Body Function. Minimally Clinically Important Difference (MCID) 5.0 and 6.2 (kg) for the affected dominant and non-dominant sides.
Motor Activity Log (MAL) | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures. The MAL is a semi-structured interview to assess arm function. ICF Domain Activity Participation. Minimal Detectable Change (MDC)MDC= 0.56- 1.06
Stroke Impact Scale (SIS). To assess physical function following stroke. ICF Domain Activity. Minimal Detectable Change (MDC)MDC >= 8 | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures
Funcitonal Independence Measure (FIM) | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures. Provides a uniform system of measurement for disability based on the International Classification of Impairment, Disabilities and Handicaps; measures the level of a patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living.ICF Domain Activity. Minimally Clinically Important Difference (MCID) FIM Total Score = 22 points
Canadian Occupational Performance Measure (COPM) | Assessments occur at baseline, 4 weeks of intervention, and at 1 month after intervention commencement.
  Secondary Outcome Measures. The COPM assesses an individual's perceived occupational performance in the areas of self-care, productivity, and leisure.ICF Domain Participation.Minimal Detectable Change (MDC) MDC for performance=1.7 points MDC for satisfaction=2.7 points

OTHER OUTCOMES:
Montreal Cognitive Assesment (MOCA) | Prior to the baseline assessment
  Exclusion criterio. Rapid screen of cognitive abilities designed to detect mild cognitive dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No